CLINICAL TRIAL: NCT04204681
Title: Tonsillar Retractor-induced Subacute Submassive Tongue Edema: A New Cause of Late Respiratory Complications in Pediatric Patients Undergoing Tonsillectomy and a Condition Detected by Ultrasonography
Brief Title: Tonsillar Retractor-induced Subacute Submassive Tongue Edema
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Professor, Selcuk University
Other Study IDs: 2018/335
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Side Effects; Tonsil Hypertrophy; Children, Only
Keywords: ultrasonography; children; tonsil; diagnostic imaging
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Patients aged 16 years or younger who were to undergo tonsillectomy surgery were eligible for inclusion in this group. Tongue areas were measured twice by submental USG.The first measurements (TA2) were done immediately after endotracheal intubation but before insertion and placement of the tonsillar retractor. The second measurements (TA1) were done after tonsillectomy surgery and after removal of the tonsillar retractor but just before extubation. The difference between TA2 and TA1 (i.e., (TA2-TA1) was used to defined the occurrence of tongue edema.
  Interventions: Diagnostic Test: Ultrasonography imaging
- Control: This group included patients aged 16 years or younger who did not need tonsillectomy surgery and any head and neck procedures. Tongue areas of the patients were measured twice by submental USG as in the study group. TA1s were done immediately after endotracheal intubation, and TA2s were done at the end of the surgical procedure just before extubation. The difference between TA2 and TA1 (i.e., (TA2-TA1) was used to defined the occurrence of tongue edema.
  Interventions: Diagnostic Test: Ultrasonography imaging

INTERVENTIONS:
Diagnostic Test: Ultrasonography imaging — This study aimed to measure the tongue areas of the patients two times both of study and control groups with ultrasonography imaging to compare the tongue areas.

SUMMARY:
This study aimed to detect tongue edema induced by the pressure exerted by tonsillar retractor; edema detection was made through tongue area measurement using ultrasonography (USG) in pediatric patients who underwent tonsillectomy surgeries.

DETAILED DESCRIPTION:
The tongue is an ideal organ for ultrasonography (USG) evaluation. This study aimed to detect the occurrence of tongue edema through USG examination and to educate clinicians about the association between subacute tongue edema and tonsillar retractor in pediatric patients.

ELIGIBILITY:
Inclusion Criteria for study group:

* Patients aged 16 years or younger
* Undergo tonsillectomy surgery
* Patients informed consent obtained from the parents

Exclusion Criteria for study group:

* Patients aged older than 16 years
* Patients with a history of syndromal craniofacial abnormalities
* Patients with systemic disorders and other otolaryngologic problems

Inclusion Criteria for control group:

* Patients aged 16 years or younger
* Patients who did not need tonsillectomy surgery and any head and neck procedures
* Patients who underwent endotracheal intubation under general anesthesia except tonsillectomy and head and neck surgery.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 16 years or younger who were to undergo tonsillectomy surgery were eligible for inclusion in this group. Informed consent was obtained from the parents of all the patients with a clinical diagnosis of chronic tonsillitis and tonsillar hypertrophy (except adenoidectomy surgeries) and were to undergo tonsillectomy surgery.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change from preoperative measurement to postoperative measurement in tongue area on the ultrasonography imaging. | 2018-2019 (6 months)
  This study aimed to evaluate the change from baseline in tongue area on the ultrasonography imaging due to the tonsillar retractor.

SECONDARY OUTCOMES:
Detection of edema formation in tongue by using ultrasonography imaging. | 2018-2019 (6 months)
  This study aimed to measure and detect the tongue edema by using ultrasonography imaging due to the tonsillar retractor.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No